CLINICAL TRIAL: NCT04447339
Title: A Retrospective, Multicenter Study of Open Nipple Sparing Mastectomy (NSM)
Brief Title: Open Nipple Sparing Mastectomy (NSM)
Acronym: NSM Open
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-RoNSM-01
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Nipple Sparing Mastectomy
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open: Prophylactic NSM cases by Open approach
  Interventions: Procedure: Nipple Sparing Mastectomy

INTERVENTIONS:
Procedure: Nipple Sparing Mastectomy — Prophylactic open NSM procedures

SUMMARY:
This is retrospective, multicenter chart review is to evaluate the complication rates of prophylactic open NSM procedures through 42 days postoperatively

DETAILED DESCRIPTION:
This is retrospective, multicenter chart review is to evaluate the complication rates of prophylactic open NSM procedures through 42 days postoperatively

ELIGIBILITY:
Inclusion Criteria:

All female patients that have undergone open prophylactic NSM cases performed between January 1, 2018 through 42 days prior to IRB approval

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Consecutive subjects that have undergone open NSM procedures for prophylaxis between January 1 2018 through 42 days prior to IRB approval will be included in this retrospective chart review.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint: complication rate | IntraOperative period through 42 days postoperatively
  To assess the number of open prophylactic nipple sparing mastectomy complications compared to the number of procedures
Effectiveness | IntraOperative period through 42 days postoperatively
  Ability to completely excise memory gland tissue and preserve Nipple Areola Complex

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - NorthShore University Health System, Evanston, Illinois
  - Mayo Clinic Hosp - Methodist Campus - MN, Rochester, Minnesota
  - Northwell Health, Queens, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Univ. of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided